CLINICAL TRIAL: NCT00073931
Title: A Phase II Trial Evaluating: Radioiodinated Anti-B1 (Anti-CD20) Antibody With Autologous Stem Cell Transplantation For Relapsed Or Refractory Non-Hodgkin's Lymphoma In Patients 60 Years Of Age And Older
Brief Title: Iodine I 131 Tositumomab Followed by Autologous Stem Cell Transplantation in Treating Older Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1366.00; CDR0000341125 (Registry Identifier: PDQ)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Peripheral Blood Stem Cell Transplantation; tositumomab I-131

INTERVENTIONS:
Biological: filgrastim — 5 µg/kg/day subcutaneously
  Other Names: G-CSF
Biological: sargramostim — 250µg/m2/d subcutaneously
  Other Names: GM-CSF
Procedure: autologous bone marrow transplantation — autologous stem cells given via central catheter
Procedure: peripheral blood stem cell transplantation — autologous stem cells given via central catheter
Radiation: tositumomab and iodine I 131 tositumomab — given intravenously (test dose of 1.7-10 mg/kg tositumomab antibody radiolabeled with ~10 mCi I-131) or via central catheter (therapy dose of 1.7-10 mg/kg tositumomab radiolabeled with individually calculated therapy dose of I-131)

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as iodine I 131 tositumomab, can locate cancer cells and deliver radioactive cancer-killing substances to them without harming normal cells. Combining a radiolabeled monoclonal antibody with autologous stem cell transplantation may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: Phase II trial to study the effectiveness of combining iodine I 131 tositumomab with autologous stem cell transplantation in treating older patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of older patients with relapsed or refractory non-Hodgkin's lymphoma treated with iodine I 131 tositumomab followed by autologous stem cell transplantation.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the toxicity and tolerability of this regimen in these patients.

OUTLINE:

* Radioimmunotherapy: Patients receive a test dose of iodine I 131 tositumomab on day -24 to determine biodistribution. Patients then receive therapeutic iodine I 131 tositumomab IV over 1 hour on day -14 and are entered into radiation isolation until day -4.
* Autologous stem cell transplantation: Patients undergo autologous bone marrow or peripheral blood stem cell transplantation on day 0. Patients undergoing bone marrow transplantation receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning on day 0 and continuing until blood counts recover.

Patients are followed at 1, 3, 6, and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 24-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma
* CD20+ disease
* Failed at least 1 prior standard systemic therapy
* Persistent lymphoma by physical examination, radiographic studies, bone marrow evaluations, flow cytometry, or polymerase chain reaction
* Tumor burden less than 500 cc by computed tomography or MRI

  * No splenomegaly
* Autologous hematopoietic stem cells or bone marrow harvested and cryopreserved

  * No circulating lymphoma cells by morphology or flow cytometry at or near the time of peripheral blood stem cell (PBSC) collection if unpurged PBSCs are to be used
  * 10% or less marrow involvement by flow cytometry or morphology if purged bone marrow is to be used
* No CNS lymphoma
* No chronic lymphocytic leukemia or small lymphocytic lymphoma/well-differentiated lymphocytic lymphoma

PATIENT CHARACTERISTICS:

Age

* 60 to 80

Performance status

* SWOG 0-1

Life expectancy

* More than 60 days

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin less than 1.5 mg/dL

Renal

* Creatinine less than 2.0 mg/dL

Cardiovascular

* No active coronary artery disease

Pulmonary

* FEV_1 at least 70% of expected
* Vital capacity at least 70% of expected

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Able to perform self-care during radiation isolation
* No major organ dysfunction
* No major infection
* No circulating anti-mouse antibody
* No other serious medical condition considered to represent contraindications to bone marrow transplantation
* No competing causes of death that would predict life span to be less than 10 additional years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior bone marrow or stem cell transplantation

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy greater than 20 Gy to any critical normal organ (e.g., lung, liver, spinal cord, or more than 25% of red marrow)

Surgery

* Not specified

Other

* More than 30 days since prior systemic antilymphoma therapy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-10; Primary Completion 2007-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Disease-free survival measured continuously | from date of transplant through date of death

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K. Gopal, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Gopal AK, Rajendran JG, Gooley TA, Pagel JM, Fisher DR, Petersdorf SH, Maloney DG, Eary JF, Appelbaum FR, Press OW. High-dose [131I]tositumomab (anti-CD20) radioimmunotherapy and autologous hematopoietic stem-cell transplantation for adults > or = 60 years old with relapsed or refractory B-cell lymphoma. J Clin Oncol. 2007 Apr 10;25(11):1396-402. doi: 10.1200/JCO.2006.09.1215. Epub 2007 Feb 20. PMID 17312330